CLINICAL TRIAL: NCT01241864
Title: Islet Transplantation in Type 1 Diabetic Kidney Allograft
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-479-A; BB-IND 11228
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogenic islet cells (human, U. Chicago) (Experimental)
  Interventions: Biological: Allogenic islet cells (human, U. Chicago); Procedure: Intraportal infusion of islet cells

INTERVENTIONS:
Biological: Allogenic islet cells (human, U. Chicago) — Human allogenic islet cells. Immunosuppression varies but may include prograf, cellcept, sirolimus, prednisone. Dosage will vary per patient based on weight. Patients will receive immunosuppression medications while islet cells are functioning.
Procedure: Intraportal infusion of islet cells — Intraportal infusion of islet cell through the portal vein in the liver.

SUMMARY:
The purpose of this study is to learn about the safety of islet transplantation when performed after kidney transplantation, which may provide more normal control of blood sugar without the need for insulin shots. Islets are special clusters of cells within the pancreas that produce insulin. These cells will be obtained from cadaver (non-living) donors and given to subjects by vein.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 to 68 years.
* Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
* Clinical history compatible with T1D with disease onset < 40 years of age and insulin-dependence for > 5 years at the time of enrollment, and a sum of subject age and insulin dependent diabetes duration of > 28.
* Absent stimulated c-peptide (< 0.3 ng/mL) in response to a MMTT [Boost® 6 mL/kg body weight (BW) to a maximum of 360 mL; another product with equivalent caloric and nutrient content may be substituted for Boost®] measured at 60 and 90 min after start of consumption.
* Subjects who are > or at 3 months post-renal transplant who are taking appropriate calcineurin inhibitor (CNI) based maintenance immunosuppression ([tacrolimus alone or in conjunction with sirolimus, mycophenolate mofetil, myfortic, or azathioprine; or cyclosporine in conjunction with sirolimus, mycophenolate mofetil, or myfortic] ± Prednisone < 10 mg/day)or subject will receive islets transplant within 72hours after kidney transplantation (islets and kidney are from the same donor)
* Stable renal function as defined by a creatinine of no more than one third greater than the average creatinine determination performed in the 3 previous months prior to islet transplantation, until rejection, obstruction or infection is ruled out.

Exclusion Criteria:

* Weight more than 90 kg or body mass index (BMI) > 30 kg/m2.
* Insulin requirement of >1.0 IU/kg/day or <15 U/day.
* Other (non-kidney) organ transplants except prior failed pancreatic graft where the graft failed within the first two weeks due to thrombosis, followed by pancreatectomy; with the pancreas transplant occurring more than 6 months prior to enrollment.
* Untreated or unstable proliferative diabetic retinopathy.
* Blood Pressure: SBP > 160 mmHg or DBP >100 mmHg despite treatment with antihypertensive agents.
* Calculated GFR < 40 mL/min/1.73 m2 using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [1]. Strict vegetarians (vegans) will be excluded only if their estimated GFR is < 35 mL/min/1.73 m2
* Proteinuria (albumin/ creatinine ratio or ACr > 300mg/g) of new onset since kidney transplantation.
* Either Class I or Class II panel-reactive anti-HLA antibodies > 50%. Subjects with either Class I or Class II panel reactive anti-HLA antibodies >50% will be excluded if any of the following are detected: Positive cross-match, Islet donor-directed anti-HLA antibodies detected by Luminex Single Antigen/specificity bead assay including weakly reactive antibodies that would not be detected by a flow cross-match, or Antibodies to the renal donor (i.e. presumed de novo).
* For female subjects: Positive pregnancy test, presently breast-feeding, desires to be pregnant at any time point in the future, which includes during or after the completion of the study even if study participation is ended early, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HbAlc <6.5% and an absence of severe hypoglycemic events | 1 year after transplantation
  The proportion of subjects with both an HbAlc <6.5% and an absence of severe hypoglycemic events at 1 year after the first islet transplant or a reduction in HbAlc of at least 1 point and an absence of severe hypoglycemic events at 1 year after the first islet transplant.

SECONDARY OUTCOMES:
HbAlc < 6.5% and an absence of severe hypoglycemic events measured after last transplant | 365 ± 14 days after the last islet transplant
  The primary endpoint measured at one year after the last islet transplant. That is the proportion of subjects with both an HbAlc < 6.5% and an absence of severe hypoglycemic events at 1 year after the last islet transplant or a reduction in HbAlc of 1 point and an absence of severe hypoglycemia at 1 year after the last islet transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Pathak P, Thampy R, Schat R, Bellin M, Beilman G, Hosseini N, Spilseth B. Transplantation for type 1 diabetes: radiologist's primer on islet, pancreas and pancreas-kidney transplantation imaging. Abdom Radiol (NY). 2024 Oct;49(10):3637-3665. doi: 10.1007/s00261-024-04368-8. Epub 2024 May 28. PMID 38806704
- [Background] Gariani K, Peloso A, Galani V, Haidar F, Wassmer CH, Kumar R, Lacin EH, Olivier V, Prada P, Compagnon P, Berishvili E, Berney T. Effect of islet alone or islets after kidney transplantation on quality of life in type 1 diabetes: A systematic review. Transplant Rev (Orlando). 2024 Dec;38(4):100870. doi: 10.1016/j.trre.2024.100870. Epub 2024 Jun 21. PMID 38917621